CLINICAL TRIAL: NCT06555874
Title: Evaluation of the MORENO Score for the Regulation of Secondary Transfers to the UAS-SMUR in Brest in Finistère in 2020
Brief Title: Evaluation of the MORENO Score for the Regulation
Acronym: ESMORTSAB19
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0075
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: the Safety / Feasibility /MORENO Score/Regulation / Secondary Transfers / SAMU 29 / Current Practices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this work is therefore to evaluate the safety and feasibility of the MORENO score for the regulation of secondary transfers to the SAMU 29 compared to current practices.

DETAILED DESCRIPTION:
Today, there is an increase in the number of secondary transfers and paramedical transport between the different hospitals in a territory. They have been promoted by the SFMU (French Society of Emergency Medicine) since 2012.

The sharp increase in the number of calls for SAMU regulation means that decisions must be made quickly and safely regarding transport requiring or not requiring a medical presence. The development of a decision support tool for the level of medicalisation of a transfer therefore seems necessary. However, there is currently no recommendation in France.

The MORENO score has already been used in a hospital in the Var, as well as in Spain and Greece. Prior validation of this score in our health territory is essential before setting up an operational procedure. Using a list of simple clinical items, this score enables us to assess whether or not it is necessary to medicalise a transfer.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients having benefited from a transfer regulated by the SAMU 29 of adult patients on the Finistère territory over a predefined period of time

Exclusion Criteria:

* Pediatric patient transfers
* Maritime transfers
* Transfers for which the collected information does not allow to establish the MORENO score.
* Patients under judicial protection (guardianship, curatorship,..)
* Opposition

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients having benefited from a transfer
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the concordance of the MORENO score for the regulation of secondary transfers at SAMU 29 and our current practices | 1 year
  Rate of agreement between our practices and the MORENO score strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement